CLINICAL TRIAL: NCT06746792
Title: Low Load, High Gains: Blood Flow Restriction's Impact on Quadriceps Adaptations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Mustafa Şakir Akgül, Associate professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KarabukUniSportsSciences
Record Dates: First submitted 2024-12-11; First posted 2024-12-24 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Healthy Individuals
Keywords: vascular occlusion; shear wave elastography; hypertrophy; muscle stiffness; strength
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle thickness (Experimental): Muscular hypertrophy , or muscle growth, refers to an increase in muscle mass. There are two types of muscular hypertrophy: myofibrillar, which is an increase in myofibrils, and sarcoplasmic, which is an increase in muscle glycogen storage.
  Interventions: Other: Low-load resistance exercise with blood flow restriction; Other: High-load resistance exercise
- Muscle stiffness and strength (Experimental): Muscle and tendon stiffness is defined as an internal resistance to changes in muscle and tendon shape caused by an external force. Muscle strength production takes place with the help of the elastic behavior of the muscles and tendons
  Interventions: Other: Low-load resistance exercise with blood flow restriction; Other: High-load resistance exercise

INTERVENTIONS:
Other: Low-load resistance exercise with blood flow restriction — BFR-RE group performed bilateral leg extension exercises to volitional exhaustion (90 seconds rest between sets, 30% 1RM) with BFR cuffs applied at 60% of limb occlusion pressure.
  Other Names: (BFR-RE)
Other: High-load resistance exercise — The HL-RE group performed the same exercise to volitional exhaustion (90 seconds rest between sets, 70% 1RM) without BFR cuffs.
  Other Names: (HL-RE)

SUMMARY:
Low-load resistance exercise with blood flow restriction (BFR-RE) presents a compelling alternative to high-load resistance exercise (HL-RE), particularly in scenarios where high loads are not feasible due to various limitations. Blood flow restriction exercise restricts blood flow to the working muscle, creating a state of ischemia. A significant advantage of BFR-RE lies in its capacity to stimulate muscle hypertrophy and strength adaptations using light external loads (20-30% 1RM), comparable to those achieved with high-load (HL) training programs that employ 70-85% 1RM As a result, BFR training has been increasingly adopted in both athletic performance and rehabilitation settings over the past few decades. Quadriceps strength and power are essential factors in both the advancement of athletic performance and the successful return to unrestricted sporting activity following injury. The findings of Culvenor et al.'s review strongly suggest that weakened quadriceps strength is a significant risk factor for symptomatic and functional decline in the knee during both activities of daily living and sport-recreational activities. Numerous electromyographic (EMG) findings suggest that single-joint and multijoint exercises elicit varying muscle activation patterns. For instance, single-joint exercises targeting the quadriceps, such as leg extensions, demonstrate higher EMG amplitudes compared to multijoint lower-extremity exercises like leg presses and squats. Resistance training, characterized by the application of high mechanical tension, remains the cornerstone for promoting muscle hypertrophy, So, research suggests that higher training intensities are associated with greater hypertrophy, up to a certain point. While both light and heavy loads have been shown to elicit similar muscle growth when sets are taken to failure. Studies have reported that high-repetition training with light loads leads to greater central fatigue. Existing literature comparing the effects of BFR-RE and HL-RE primarily focuses on the some quadriceps and hamstring muscle group and its associated exercises. However, none of these studies employed a training protocol in which sets were taken to or near failure.

ELIGIBILITY:
Inclusion Criteria:

* keep healthy
* must be able to attend training regularly

Exclusion Criteria:

* smoking habit
* had orthopedic conditions that hindered lower-body resistance exercise, had hypertension (140/90 mm Hg), or had a BMI exceeding 30 kg/m2

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-03-29 (Estimated); Study Completion 2025-03-29 (Estimated)

PRIMARY OUTCOMES:
Thigh Circumference | 2 day
  Measurement of thigh circumference was performed at a point 33% distal to the inguinal crease, precisely matching the intended cuff application site as verified by a trained investigator. The inguinal crease-to-superior patellar pole distance was also recorded using a standard anthropometric tape measure
Muscle Strength Test | 2 day
  Prior to commencing the strength assessment, using a Lafayette Manual Muscle Testing System (Lafayette Instrument Company, Lafayette®) a period of familiarization was allowed between the examiner and participant. Subsequently, a trained examiner guided the participant through a series of practice repetitions of leg flexion, and leg extension movements until correct execution was confirmed. The order of movements was randomized. The participant was then verbally instructed to perform three maximal contractions for each movement (3-second hold). A 1-minute rest interval was incorporated between successive contractions, and a 3-minute rest interval was implemented between different movement sets. Measurement of leg extension were obtained with participants in a seated position, while leg flexion measurement were taken with participants in a prone position.
Muscle Thickness Assessment | 4 day
  Subjects had not engaged in physical activity before the study (48-72 hours), and muscle thickness (MT) was measured at a prone rest position. All muscle thickness measurements were obtained with a single ultrasound device equipped with a 2-9 MHz linear transducer. A researcher (medical doctor, N.K.K) who was blinded to the exercise groups with more than 10 years of experience in musculoskeletal imaging performed all measurement
Muscle Stiffness and Shear Wave Elastography | 4 day
  After the muscle thickness measurements, the stiffness measurements of quadriceps muscle were obtained using the shear wave elastography (SWE) imaging option of the same ultrasound device with the same linear transducer.

OTHER OUTCOMES:
Anthropometric Measurements | One day
  Height, weight and Body mass index (BMI) were measured using a stadiometer (InBody 270 (Biospace, California, USA), with subjects wearing light clothing and no shoes. Measurements were taken before the exercise program.
Blood Pressure | One day
  After a 5-minute supine rest, participants' left brachial blood pressure (BP) was measured twice (1-minute interval). The average of the two closest readings (within 5 mmHg) was recorded in mmHg
Heart Rate | One day
  After a 5-minute supine rest

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk University Faculty of Sports Sciences, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All antropometric and muscle strength, muscle thickness, and muscle stiffness parameters will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR